CLINICAL TRIAL: NCT03941184
Title: Determining the Association Between Spontaneous Coronary Artery Dissection (SCAD) and Autoimmunity
Brief Title: Spontaneous Coronary Artery Dissection (SCAD) and Autoimmunity
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marysia Tweet, Principal Investigator, Mayo Clinic
Other Study IDs: 19-002489
Record Dates: First submitted 2019-04-01; First posted 2019-05-07 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: SCAD; Addison Disease; Ankylosing Spondylitis; Antiphospholipid Antibody Syndrome; Celiac Disease; Crohn Disease; Dermatomyositis; Polymyositis; Guillain-Barre Syndrome; Hepatitis, Autoimmune; Graves Disease; Hashimoto Thyroiditis; Multiple Sclerosis; Myasthenia Gravis; Pernicious Anemia; Polymyalgia Rheumatica; Primary Biliary Cirrhosis; Psoriasis; Rheumatoid Arthritis; Systemic Sclerosis; Sjögren Syndrome; Systemic Lupus Erythematosus; Takayasu Arteritis; Type 1 Diabetes Mellitus; Ulcerative Colitis; Uveitis; Vasculitis; Vitiligo; Raynaud
Keywords: spontaneous coronary artery dissection; autoimmune; incidence
MeSH Terms: conditions — Addison Disease; Spondylitis, Ankylosing; Antiphospholipid Syndrome; Celiac Disease; Crohn Disease; Dermatomyositis; Polymyositis; Guillain-Barre Syndrome; Hepatitis, Autoimmune; Graves Disease; Hashimoto Disease; Multiple Sclerosis; Myasthenia Gravis; Anemia, Pernicious; Polymyalgia Rheumatica; Liver Cirrhosis, Biliary; Psoriasis; Arthritis, Rheumatoid; Scleroderma, Systemic; Sjogren's Syndrome; Lupus Erythematosus, Systemic; Takayasu Arteritis; Diabetes Mellitus, Type 1; Colitis, Ulcerative; Uveitis; Vasculitis; Vitiligo; Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCAD cases: SCAD cases will be identified based on presence of at least one diagnosis code for SCAD followed by manual verification by a trained individual, OR, inclusion in the previously validated SCAD cohort (Tweet 2012).
- Controls without SCAD: Potential controls will be identified based on absence of any SCAD diagnosis codes.

SUMMARY:
This case control study aims to determine whether spontaneous coronary artery dissection (SCAD) is associated with autoimmune diseases and to update the incidence of SCAD in a population-based cohort.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 110
* Residence in Olmsted County. Note: if sufficient numbers cannot be reached using only Olmsted County, will expand to the 27-county region.

Exclusion Criteria:

* None

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Rochester Epidemiology Project (REP) is a population-based cohort that includes medical record data for over 500,000 unique individuals who resided in Olmsted County at some point between 1966 and the present, and received health care for any reason within the system (St. Sauver 2012).
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 1995-01-01 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Odds of autoimmune disease in SCAD cases compared to controls | Through study completion, or approximately 50 years (average age of study participants)
Incidence Rate of SCAD | Through study completion, or approximately 50 years (average age of study participants)

SECONDARY OUTCOMES:
SCAD recurrence | Through study completion, or approximately 50 years (average age of study participants)

OTHER OUTCOMES:
Odds of laboratory markers for autoimmune disease in SCAD cases compared to controls | Through study completion, or approximately 50 years (average age of study participants)
Odds of validated rheumatoid arthritis in SCAD cases compared to controls | Through study completion, or approximately 50 years (average age of study participants)
  using the Rochester Epidemiology Project Rheumatoid Arthritis cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tweet MS, Hayes SN, Pitta SR, Simari RD, Lerman A, Lennon RJ, Gersh BJ, Khambatta S, Best PJ, Rihal CS, Gulati R. Clinical features, management, and prognosis of spontaneous coronary artery dissection. Circulation. 2012 Jul 31;126(5):579-88. doi: 10.1161/CIRCULATIONAHA.112.105718. Epub 2012 Jul 16. PMID 22800851
- [Background] McGonagle D, McDermott MF. A proposed classification of the immunological diseases. PLoS Med. 2006 Aug;3(8):e297. doi: 10.1371/journal.pmed.0030297. PMID 16942393
- [Background] St Sauver JL, Grossardt BR, Yawn BP, Melton LJ 3rd, Pankratz JJ, Brue SM, Rocca WA. Data resource profile: the Rochester Epidemiology Project (REP) medical records-linkage system. Int J Epidemiol. 2012 Dec;41(6):1614-24. doi: 10.1093/ije/dys195. Epub 2012 Nov 18. PMID 23159830
- [Background] Tweet MS, Kok SN, Hayes SN. Spontaneous coronary artery dissection in women: What is known and what is yet to be understood. Clin Cardiol. 2018 Feb;41(2):203-210. doi: 10.1002/clc.22909. Epub 2018 Mar 1. PMID 29493808
- [Background] Hayes SN, Kim ESH, Saw J, Adlam D, Arslanian-Engoren C, Economy KE, Ganesh SK, Gulati R, Lindsay ME, Mieres JH, Naderi S, Shah S, Thaler DE, Tweet MS, Wood MJ; American Heart Association Council on Peripheral Vascular Disease; Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Genomic and Precision Medicine; and Stroke Council. Spontaneous Coronary Artery Dissection: Current State of the Science: A Scientific Statement From the American Heart Association. Circulation. 2018 May 8;137(19):e523-e557. doi: 10.1161/CIR.0000000000000564. Epub 2018 Feb 22. PMID 29472380
- [Background] Adlam D, Alfonso F, Maas A, Vrints C; Writing Committee. European Society of Cardiology, acute cardiovascular care association, SCAD study group: a position paper on spontaneous coronary artery dissection. Eur Heart J. 2018 Sep 21;39(36):3353-3368. doi: 10.1093/eurheartj/ehy080. No abstract available. PMID 29481627
- [Background] Waterbury TM, Tweet MS, Hayes SN, Eleid MF, Bell MR, Lerman A, Singh M, Best PJM, Lewis BR, Rihal CS, Gersh BJ, Gulati R. Early Natural History of Spontaneous Coronary Artery Dissection. Circ Cardiovasc Interv. 2018 Sep;11(9):e006772. doi: 10.1161/CIRCINTERVENTIONS.118.006772. PMID 30354594
- [Background] Tweet MS, Eleid MF, Best PJ, Lennon RJ, Lerman A, Rihal CS, Holmes DR Jr, Hayes SN, Gulati R. Spontaneous coronary artery dissection: revascularization versus conservative therapy. Circ Cardiovasc Interv. 2014 Dec;7(6):777-86. doi: 10.1161/CIRCINTERVENTIONS.114.001659. Epub 2014 Nov 18. PMID 25406203
- [Background] Tweet MS, Hayes SN, Codsi E, Gulati R, Rose CH, Best PJM. Spontaneous Coronary Artery Dissection Associated With Pregnancy. J Am Coll Cardiol. 2017 Jul 25;70(4):426-435. doi: 10.1016/j.jacc.2017.05.055. PMID 28728686
- See also: The "Virtual" Multicenter Spontaneous Coronary Artery Dissection (SCAD) Registry — https://clinicaltrials.gov/ct2/show/NCT01429727
- See also: Genetic Investigations in Spontaneous Coronary Artery Dissection (SCAD) — https://clinicaltrials.gov/ct2/show/NCT01427179